CLINICAL TRIAL: NCT02917590
Title: Dual Task Obstacle Crossing: Effects on Walking and Balance Ability, and Relationship With Falls in Independent Ambulatory Patients With Spinal Cord Injury
Brief Title: Dual-task Obstacle Crossing Training in Ambulatory Subjects With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Khon Kaen University (Other)
Responsible Party: Principal Investigator, Sugalya Amatachaya, Assoc. Prof. Dr, Khon Kaen University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: PHD/0128/2556
Record Dates: First submitted 2016-09-22; First posted 2016-09-28 (Estimated); Last update posted 2016-09-28 (Estimated); Status verified 2016-09

CONDITIONS: Injuries, Spinal Cord
Keywords: Spinal cord injury; dual-task obstacle crossing
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dual-task obstacle crossing training (Experimental): The four obstacles in the sizes of 4cm wide, 8cm wide, 4cm high, and 8cm high are randomly placed along a 10-meter walkway in 2-meter intervals. Subjects are instructed to walk continuously over obstacles at their comfortable speed, as good as they can without contact the obstacles by their leg or device. During walk over obstacles, subjects asked to perform simultaneously with a color word stroop task which requires subjects to see and answer the color of the name of a color words in the monitor (ignore the meaning) as quickly as possible, and loudly.
  Interventions: Other: Dual-task obstacle crossing training
- Single-task obstacle crossing training (Sham Comparator): The four obstacles in the sizes of 4cm wide, 8cm wide, 4cm high, and 8cm high are randomly placed along a 10-meter walkway in 2-meter intervals. Subjects are asked to walk continuously over obstacles at their comfortable speed, as good as they can without contact the obstacles by their leg or device.
  Interventions: Other: Single-task obstacle crossing training

INTERVENTIONS:
Other: Dual-task obstacle crossing training — Obstacle crossing simultaneously a color word stroop task training
  Arms: Dual-task obstacle crossing training
Other: Single-task obstacle crossing training — Obstacle crossing training
  Arms: Single-task obstacle crossing training

SUMMARY:
Is dual-task obstacle crossing training more efficiently than single-task obstacle crossing training on the improvement of walking ability, balance ability, and lower extremity muscle strength in ambulatory subjects with spinal cord injury

DETAILED DESCRIPTION:
To compare immediate effects of dual-task and single-task obstacle crossing training in ambulatory subjects with spinal cord injury

ELIGIBILITY:
Inclusion Criteria:

* independent ambulatory subjects with
* traumatic causes or non-progressive diseases
* sub-acute and chronic stage of injury (at least 3 month after injury)
* body mass index (BMI) between 18.5-29.9 kg/m2
* walk independently for at least 17 meters with or without assistive devices (Functional Independence Measure Locomotor (FIM-L) scores 5-7)
* able to read Thai

Exclusion Criteria:

* pain in the musculoskeletal system with a pain scale more than 5 out of 10 on a the visual analog scale (VAS)
* deformity in the joints that affect ambulatory ability
* unable to understand the commands and tests used in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 7 (Actual)
Dates: Start 2015-10; Primary Completion 2017-02 (Estimated); Study Completion 2017-07 (Estimated)

PRIMARY OUTCOMES:
10MWT (Single-task) | 1 day
  Walking speed in single-task condition

SECONDARY OUTCOMES:
10MWT (Dual-task) | 1 day
  Walking speed in dual-task condition
TUGT | 1 day
  Balance ability
FTSST | 1 day
  Lower extremity muscle strength

CONTACTS AND LOCATIONS:
Overall Officials: Sugalya Amatachaya, PhD, Principal Investigator — School of Physical Therapy, Faculty of Associated Medical Sciences, Khon Kaen University, Thailand

IPD SHARING:
Plan to Share IPD: No